CLINICAL TRIAL: NCT03745001
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Food Effect of Single Ascending Doses and Multiple Ascending Doses of EHP-101 in Healthy Subjects
Brief Title: To Evaluate the Safety and Tolerability, Pharmacokinetics, Food-effect and Pharmacodynamics of EHP-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emerald Health Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EHP-101-01
Record Dates: First submitted 2018-10-03; First posted 2018-11-19 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study
Who Masked: Participant, Investigator
Masking Description: EHP-101 Liquid or matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single dose study part (Experimental): there will be 7 cohorts of healthy volunteers dosed with single doses of EHP-101 (7 planned dose levels) or with placebo and 1 potential additional cohort (also dosed with single dose of EHP-101 or placebo)
  Interventions: Drug: EHP-101 Liquid single dose; Drug: Matching placebo
- Multiple dose study part (Experimental): there will be 3 cohorts of healthy volunteers dosed with multiple doses of EHP-101 (3 planned dose levels) or placebo and 1 potential additional cohort (also dosed with multiple doses of EHP-101 or placebo)
  Interventions: Drug: EHP-101 Liquid multiple doses; Drug: Matching placebo

INTERVENTIONS:
Drug: EHP-101 Liquid single dose — One single oral administration with EHP-101 liquid formulation. The doses will be ascending per cohort from 0.91 mg to 200 mg. The initially planned once daily dose regimen may be modified by the Safety Review Committee based on emerging PK data, eg, assigned dose levels may be divided into 2 doses administered 12 hours apart (twice a day).
  Arms: Single dose study part
Drug: EHP-101 Liquid multiple doses — One single daily administration with EHP-101 liquid formulation during 7 consecutive days. The doses will be ascending per cohort. Each ascending level will not exceed the tested dose levels in the single dose part of the study. The initially planned once daily dose regimen may be modified by the Safety Review Committee based on emerging PK data, eg, assigned dose levels may be divided into 2 doses administered 12 hours apart (twice a day)
  Arms: Multiple dose study part
Drug: Matching placebo — Oral liquid administration daily

SUMMARY:
The study will assess the safety and tolerability, pharmacodynamic, pharmacokinetic profiles, and food effect of single ascending doses and multiple ascending doses (7 consecutive days) after daily oral administration in healthy male and female subjects.

DETAILED DESCRIPTION:
This Phase 1, single center, randomized, double-blind, placebo-controlled study will be conducted in 2 parts: the single ascending dosing (SAD) will constitute Part 1 and the multiple ascending dosing (MAD) will constitute Part 2. In Part 1 (ie, SAD) of the study, up to 64 eligible subjects will be randomized with an allocation ratio of 3:1 to receive EHP-101 Liquid or matching placebo within one of up to 8 sequential cohorts; Sentinel subjects (1 receiving EHP-101 Liquid and 1 receiving placebo) will be dosed prior to dosing the remaining 6 subjects to allow for observation of adverse reactions before exposing the Investigational Product (IP) to a greater number of subjects, in the SAD cohorts. In Part 2 of the study, up to 40 eligible subjects will be randomized with an allocation ratio of 4:1 to receive EHP 101 Liquid or matching placebo within one of up to 4 cohorts. Dose-escalations, initiation of a single-dose food effect cross-over investigation and the start of the MAD part of the study will be coordinated by a Safety Review Committee (SRC) following review of available safety data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects ≥ 18 to ≤ 65 years of age.
* Body mass index (BMI) range 18 to 34 kg/m².
* Free from any clinically significant abnormality on the basis of medical history, vital signs, physical examination, 12-lead electrocardiogram (ECG), echocardiography, ophthalmologic examinations and tests, and laboratory evaluations at screening and admission, as judged by the Investigator.
* Cardiac Troponin I level below the upper limit of normal, as defined by the manufacturer.
* Ability to understand and the willingness to provide informed consent for participation in the study.
* Ability and willingness, as judged by the Investigator, to comply with all study requirements.

Exclusion Criteria:

* Any known, documented, or suspected history of:

  1. schizophrenia or other psychotic illness, or diagnosis of schizophrenia in a first-degree relative.
  2. alcohol or substance abuse within the last 2 years before screening or positive test result(s) for alcohol and or drugs of abuse.
  3. Regular alcohol consumption >21 units per week
* Use of nicotine or nicotine-containing products during participation in the study.
* Caffeine consumption is limited to no more than 2 units per day.
* Any known, documented, or suspected hypersensitivity to cannabinoids or any of the excipients of EHP-101 Liquid.
* Use of cannabis or cannabinoid-based medications.
* Abnormal screening 12-lead ECG interpreted by the Investigator to be clinically significant.
* Presence of ophthalmologic abnormalities at baseline, specifically known closed angles, previous laser iridotomy, or severe hypermetropic diagnosis.
* Male subjects who are not surgically sterilized and who do not agree to use condoms in combination with partner use of a highly effective method of contraception. Female subjects of childbearing potential who are not using a highly effective method of contraception, as judged by the Investigator, and who do not consent: i) to use a combined barrier method of contraception and ii) to remain on a highly effective method of contraception while receiving study intervention during the study and for at least 90 days after the end of study treatment.
* Female subjects who are pregnant, lactating, or planning pregnancy during the course of the study and for 12 weeks thereafter.
* Male subjects unwilling to abstain from sperm donation during the study and for 12 weeks thereafter.
* Any evidence or history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV types 1 and 2) infection.
* Subjects who have received an IP within the 12 weeks before the screening visit.
* Blood donation or loss (eg, ≥ 400 mL) within 3 months before enrollment and unwilling to abstain from blood donation during the study.
* Significant disease or disorder, which, in the opinion of the Investigator or other staff who is directly involved in the study, may either put the subject at risk because of participation in the study or interfere with the subject's ability to participate in the study.
* Intake of any metabolic enzyme-affecting drugs from 30 days prior to Day -1 (ie, Check-in).
* Vaccination within 30 days prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-08-11 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) including serious adverse events (SAEs) following single and multiple ascending oral doses for 30 days after dosing. | From the time of the first dose and continued until 30 days after
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments.

SECONDARY OUTCOMES:
Time to reach VCE-004.8 maximum concentration after a single drug administration (Tmax). | Starting 1 hour prior to dosing on Day 1 and until 192 hours after dosing on Day 9.
  Serum samples will be collected on Day 1: 1 hour predose; 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours post dose, on Day 2: 24 hours post dose, on Day 3: 48 hours post dose, on Day 4: 72 hours post dose, on Day 5: 96 hours postdose, on Day 6: 120 hours postdose, on Day 7: 144 hours post dose, on Day 8, 168 hours, on Day 9: 192 hours post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above. * samples to be collected on Day 1 only for the modified dose regimen.
  In one cohort the outcome measure is done once without food intake and once after the intake of a high fat breakfast (in 2 different periods). Both outcomes (with and without breakfast intake) will be compared to assess the effect of a high fast breakfast on VCE-004.8 Tmax.
Observed maximum VCE-004.8 serum concentration following single drug administration (Cmax). | Starting 1 hour prior to dosing on Day 1 and until 192 hours after dosing on Day 9.
  Serum samples will be collected on Day 1: 1 hour predose; 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours post dose, on Day 2: 24 hours post dose, on Day 3: 48 hours post dose, on Day 4: 72 hours post dose, on Day 5: 96 hours postdose, on Day 6: 120 hours postdose, on Day 7: 144 hours post dose, on Day 8, 168 hours, on Day 9: 192 hours post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above. * samples to be collected on Day 1 only for the modified dose regimen.
  In one cohort the outcome measure is done once without food intake and once after the intake of a high fat breakfast (in 2 different periods). Both outcomes (with and without breakfast intake) will be compared to assess the effect of a high fast breakfast on VCE-004.8 Cmax.
Area under the serum VCE-004.8 concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) following single drug administration. | Starting 1 hour prior to dosing on Day 1 and until 192 hours after dosing on Day 9.
  Serum samples will be collected on Day 1: 1 hour predose; 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*, 15 hours*; 16 hours post dose, on Day 2: 24 hours post dose, on Day 3: 48 hours post dose, on Day 4: 72 hours post dose, on Day 5: 96 hours postdose, on Day 6: 120 hours postdose, on Day 7: 144 hours post dose, on Day 8, 168 hours, on Day 9: 192 hours post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 only for the modified dose regimen.
  In one cohort the outcome measure is done once without food intake and once after the intake of a high fat breakfast (in 2 different periods). Both outcomes (with and without breakfast intake) will be compared to assess the effect of a high fast breakfast on VCE-004.8 AUClast
Time to reach VCE-004.8 maximum concentration after a multiple drug administration (Tmax). | Starting 1 hour prior the first dose administration (Day 1) until 24 hours after the first dose administration on Day 7.
  Serum samples will be collected on Day 1 and Day7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*, 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose.
  This outcome measure shows the mean of all subject values resulting from each time point specified above.*samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
Time to reach VCE-004.8 maximum concentration after a multiple drug administration (Tmax). | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the last dose administration on Day 12
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose.
  This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
Observed maximum VCE-004.8 serum concentration following multiple drug administration (Cmax). | Starting 1 hour prior the first dose administration (Day 1) until 24 hours after the first dose administration on Day 8
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
Observed maximum VCE-004.8 serum concentration following drug administration at steady state (Cmax,ss) after multiple drug administration | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the first dose administration on Day 12
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
Area under the serum VCE-004.8 concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) after the first dose administration during multiple drug administration | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the first dose administration on Day 12
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
The area under the serum VCE-004.8 concentration-time curve from time zero to the end of the dosing interval tau at steady state (AUCtau,ss) during multiple drug administration | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the last dose administration on Day 12.
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
The average steady state VCE-004.8 serum concentration during multiple dosing (Cav,ss) after multiple dose administration | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the last dose administration on Day 12.
  Serum samples will be collected on Day 1: 1 hour predose; 0,25 hour; 0,5 hour; 1 hour; 1,5 hours; 2 hours; 3 hours; 4 hours; 6 hours; 8 hours; 12 hours; 14 hours*; 15 hours*; 16 hours post dose, on Day 2: 24 hours post dose, on Day 3: 1 hour prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1 hour prior dosing, on Day 15 (last time the drug is administered): 1 hour predose; 0,25 hour; 0,5 hour; 1 hour; 1,5 hours; 2 hours; 3 hours; 4 hours; 6 hours; 8 hours; 12 hours; 16 hours post dose, on Day 16: 24 hours post dose and Day 17: 48 hours post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
The effective VCE-004.8 half-life based on drug accumulation at steady state (T1/2,acc) after multiple dose administration | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the last dose administration on Day 12.
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.
The accumulation VCE-004.8 ratio (Racc) after multiple drug administration | Starting 1 hour prior the first dose administration (Day 1) until 120 hours after the last dose administration on Day 12.
  Serum samples will be collected on Day 1 and Day 7: 1 hour predose; Day 1 and 7: 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 6 hours; 9 hours; 12 hours; 14 hours*; 15 hours*; 16 hours and on Day 8: 24 hours post dose, on Day 9: 48 hours post dose, on Day 10: 72 hours post dose, on Day 11: 96 hours postdose, and on Day 12: 120 hours postdose. This outcome measure shows the mean of all subject values resulting from each time point specified above. *samples to be collected on Day 1 and Day 7 only for the modified dose regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Snyder, MD, Study Chair — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No